CLINICAL TRIAL: NCT07083115
Title: Developing MRI Technologies for Atrial Fibrillation
Status: Not yet recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Christopher Nguyen, Director of Cardiovascular Innovation Research Center, The Cleveland Clinic
Other Study IDs: 25-073
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Cardiac MRI; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To measure image quality of damaged areas of the heart in patients with Atrial fibrillation using the contrast Gadopiclenol vs conventional Gadolinium-based contrast agents(GBCA)

DETAILED DESCRIPTION:
With the use of gadolinium-based contrast agents (GBCA), cardiac MRI has become the clinical gold standard in tissue characterization of fibrosis in the ventricular myocardium. More recently, contrast enhanced cardiac MRI using standard class I GBCA was proposed to reveal fibrosis in the left atrium to characterize AF via the DECAF and DECAF II studies.

Unfortunately, the results were negative with the culprit reason being the lack of clear visualization of the enhanced regions. This claim was substantiated in a recent 2024 Langendorff (reanimated ex vivo) human heart study in AF patients showing clearly the presence of fibrosis with microscopy and more importantly it showed contrast enhanced MRI can also visualize the fibrosis an equivalent 4x dose of GBCA. However, the study was performed ex vivo and no follow up in vivo study was performed to test the in vivo viability. Thus the investigators propose the unique use of standard dose of Gadopiclenol (Elucerim), a novel high relaxivity agent, contrast enhanced MRI to scan AF patients to identify and characterize areas of fibrosis and validate the electrophysiology dysfunction in those same regions.

It is hypothesized that the Gadopiclenol can provide an improved enhancement as compared to the use of conventional GBCA like Gadovist and potentially can better reveal the AF fibrotic infiltrate. Furthermore, the higher contrast to noise ratio (CNR) of the lesion will support a significantly higher spatial resolution and potentially enable sub-mm high resolution imaging.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of Atrial Fibrillation

Exclusion Criteria:

* Contraindications to MRI
* Contraindications to Gadolinium based contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients screened for atrial fibrillation from established afib clinics
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Image quality | At completion of each MRI
  To demonstrate standard dose (0.05mmol/kg) of Gadopiclenol cardiac MRI significantly improves the enhancement of AF compared with standard dose (0.1mmol/kg) of conventional GBCA agents. Research MRI data will be reviewed against any standard clinical MRI available in the patient's medical record.

SECONDARY OUTCOMES:
High resolution Cardiac MRI for improved imaging of AF | At completion of each MRI
  To demonstrate standard dose (0.05mmol/kg) of Gadopiclenol can enable ultra-high resolution sub-mm cardiac 3D MRI scan for significantly improved imaging of AF. AF patients (N=100), will be recalled for a research scan using the proposed Gadopiclenol contrast agent. The research scan will use a novel 0.9 mm isotropic 3D LGE scan. Wall sharpness measured in units of (1/mm) and lesion CNR will be calculated for both scans and compared. Scan time for both sequences will be made equal.
  The primary outcome is in Aim 1 of comparing Gadopiclenol cardiac MRI scans with conventional GBCA cardiac MRI in the context of LA enhancement via contrast to noise ratio (CNR). Previous work in our group using a standard dose of GBCA in RF ablated pigs shows an effect size of about 1.0 in CNR between Gadopiclenol and conventional GBCA in LV enhancement. Assuming this effect size, 80% statistical power, and an alpha = 0.5, it would require at least 32 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nguyen, PhD, Principal Investigator — The Cleveland Clinic